CLINICAL TRIAL: NCT05042934
Title: Phase 1B/2 Study of Lurbinectedin With or Without Irinotecan for Patients With Relapsed or High Risk Chemotherapy-Naive Ewing Sarcoma
Brief Title: Lurbinectedin With or Without Irinotecan in Treating Patients With Relapsed or High Risk Metastatic Ewing Sarcoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI stated trial no longer fits the framework & portfolio of work that is prioritized by the department. PI will not have the anticipated accrual in PI view to complete the study. Given that, PI request this protocol be closed prior to its activation.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0607; NCI-2019-01258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0607 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-07; First posted 2021-09-13 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Ewing Sarcoma; Recurrent Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Biopsy, Fine-Needle; Irinotecan; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lurbinectedin, fine-needle aspiration, irinotecan) (Experimental): Patients receive lurbinectedin IV over 60 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo fine-needle aspiration on days 2-6 of cycle 1. Beginning in cycle 2, if the biopsy shows suppression of NR0B1, then patients receive irinotecan IV over 1 hour on the day of maximum NR0B1 suppression on cycle 2. If the duration of NR0B1 suppression from lurbinectedin alone exceeds 48 hours, or if the duration of NR0B1 suppression from lurbinectedin and irinotecan exceeds 48 hours and is longer than that seen with lurbinectedin alone, then patients may receive a second dose of irinotecan during the extended period of NR0B1 suppression.
  Interventions: Procedure: Fine-Needle Aspiration; Drug: Irinotecan; Drug: Irinotecan Hydrochloride; Drug: Lurbinectedin

INTERVENTIONS:
Procedure: Fine-Needle Aspiration — Undergo fine-needle aspiration
  Other Names: Aspirate, Fine Needle; Fine Needle Aspiration; Fine Needle Biopsy; fine-needle aspiration biopsy; FNA; FNA biopsy
Drug: Irinotecan — Given IV
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Drug: Lurbinectedin — Given IV
  Other Names: PM01183; Zepzelca

SUMMARY:
This phase Ib/II trial studies best dose and side effects of lurbinectedin and how well it works with or without irinotecan in treating patients with Ewing sarcoma that has come back (relapsed) or is high risk and has spread to other places in the body (metastatic). Lurbinectedin may decrease chemicals in the body related to Ewing sarcoma, and reducing these chemicals may make the tumor cells more sensitive to irinotecan. Chemotherapy drugs, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving lurbinectedin with or without irinotecan may work better in treating patients with Ewing sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the time course of nuclear receptor subfamily 0 group B member 1 (NR0B1) suppression, Werner syndrome RecQ like helicase (WRN) suppression, and S-phase blockade after lurbinectedin (PM01183) administration in patients with Ewing sarcoma and Ewing's Sarcoma-Friend leukemia integration 1 transcription factor (EWS-FLI1) translocation. (Phase IB) II. To determine whether similar NR0B1 suppression, and S-phase blockade after lurbinectedin (PM01183) administration is seen in patients with Ewing sarcoma other EWSR1 translocations. (Phase IB) III. To determine the recommended dose (RD) of lurbinectedin (PM01183) in combination with irinotecan every 3 weeks for patients with relapsed Ewing sarcoma. (Phase IB) IV. To assess the activity of lurbinectedin in combination with low-dose irinotecan in patients with relapsed Ewing sarcoma. (Phase II) V. To assess if the suppression of NR0B1is extended after combining irinotecan with lurbinectedin. (Phase II) VI. To assess the histological characteristics of patients with prolonged stable disease to determine if they are true responders. (Phase II)

OUTLINE: This is a phase Ib, dose-escalation study of lurbinectedin, followed by a phase II study.

Patients receive lurbinectedin intravenously (IV) over 60 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo fine-needle aspiration on days 2-6 of cycle 1. Beginning in cycle 2, if the biopsy shows suppression of NR0B1, then patients receive irinotecan IV over 1 hour on the day of maximum NR0B1 suppression on cycle 2. If the duration of NR0B1 suppression from lurbinectedin alone exceeds 48 hours, or if the duration of NR0B1 suppression from lurbinectedin and irinotecan exceeds 48 hours and is longer than that seen with lurbinectedin alone, then patients may receive a second dose of irinotecan during the extended period of NR0B1 suppression.

After completion of study treatment, patients are followed up at 30 days, every 2 months for 6 months, and then every 3 months for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Patients of any age >= 16 with documented Ewing sarcoma with disease accessible for repeated fine-needle aspiration biopsies who have relapsed after or are considered high-risk (unlikely to be cured by standard therapy) are eligible for the initial pharmacologic investigations. The previously untreated patients will be treated only with a single dose of lurbinectedin as if in a "window" protocol
* Patients must have a confirmed diagnosis of Ewing sarcoma, measurable evaluable disease, and have relapsed after standard chemotherapy or have high-risk metastatic disease unlikely to be cured with standard therapy (such as multiple bone metastases). a. Phase I: Patients must have documented Ewing sarcoma with disease accessible for repeated fine-needle aspiration biopsies. b. Phase II: Patients must have relapsed after initial curative or palliative therapy. Disease accessible for repeated biopsies is not required
* Phase II: Patients of any age >= 16 with documented Ewing sarcoma who have relapsed after initial curative or palliative therapy are eligible. Disease accessible for repeated biopsies is not required
* Patients may have any translocation type, but a sufficient number of EWS-FLI1 patients to meet objectives 1, 3, and 4 is required for study completion
* Prior treatment with irinotecan is permitted
* Estimated life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must be >= 2 weeks beyond treatment of any chemotherapy, other investigational therapy, biological, targeted agents or radiotherapy, and must have recovered to =< grade 1 toxicity or previous baseline for each toxicity
* Abnormal organ function is permitted
* Absolute neutrophil count >= 1500/mL
* Platelets >= 100,000/mL unless due to bone-marrow infiltration by tumor
* Creatinine =< 1.5 x upper limit of normal (ULN) (or calculated glomerular filtration rate [GFR] > 30 ml/min)
* Bilirubin =< 1.6 mg/dL (1.5 x ULN) or direct bilirubin =< 0.3 mg/dL
* Aspartate transaminase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and/or alanine transaminase (ALT)/serum glutamic-pyruvic transaminase (SGPT) =< 2.5 x upper limit of normal (ULN)
* International normalized ratio (INR) =< 2
* Albumin >= 3.0 g/dL
* Women of childbearing potential (WOCBP) MUST have a negative serum or urine human chorionic gonadotropin (hCG) test unless prior hysterectomy or menopause (defined as 12 consecutive months without menstrual activity). Patients should not become pregnant or breastfeed while on this study. Sexually active patients must agree to use contraception prior to study entry, for the duration of study participation, and for 3 months after the last dose. Highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  * Total abstinence or male/female sterilization
* During Phase 1, the multiple fine needle aspirations must be safe and feasible, and patients must consent to the performance of those multiple fine needle aspirations
* Signed informed consent obtained prior to any screening procedures

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients who are pregnant or breastfeeding
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 6 months after the end of treatment
* Patients with uncontrolled intercurrent illness including, but not limited to active infection requiring hospitalization
* Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B virus surface antigen [Hbs/Ag], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA])
* Active, bleeding diathesis
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Prior treatment with PM01183, or trabectedin
* Evident symptomatic pulmonary fibrosis or interstitial pneumonitis, pleural or cardiac effusion rapidly increasing and/or necessitating prompt local treatment within seven days
* Known hypersensitivity to irinotecan

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Time course of nuclear receptor subfamily 0 group B member 1 (NR0B1) suppression, Werner syndrome RecQ like helicase (WRN) suppression, and S-phase blockade (Phase IB) | Up to 2 years
  All analyses of data will be descriptive in nature.
NR0B1 suppression, and S-phase blockade after lurbinectedin (Phase IB) | Up to 2 years
  All analyses of data will be descriptive in nature.
Recommended dose of lurbinectedin (Phase IB) | Up to 21 days
  Dose-limiting toxicity is defined as grade 3 or 4 toxicity that does not resolve to grade 1 or less by 4 weeks.
Suppression extension of NR0B1 (Phase II) | Up to 2 years
Histological characteristics of patients (Phase II) | Up to 2 years
  Will assess the histological characteristics of patients to determine if they are true responders by descriptive statistics.
Progression-free survival (PFS) (Phase II) | Time from treatment onset to either disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) or death from any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted on PFS. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Overall survival (OS) (Phase II) | Time from treatment onset to death, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted on OS. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure that the models are appropriate.
Overall response rate (Phase II) | At 6 weeks
  Will be defined as evidence of complete or partial response 6 weeks after the initiation of combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Benjamin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org